CLINICAL TRIAL: NCT00915525
Title: Long Term Follow-up Study of Safety and Efficacy of Botulinum Toxin Type A for the Treatment of Patients With Idiopathic Overactive Bladder With Urinary Incontinence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 191622-096
Record Dates: First submitted 2009-05-28; First posted 2009-06-08 (Estimated); Results first posted 2015-12-18 (Estimated); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Overactive Bladder; Urinary Incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- botulinum toxin Type A 100U (Experimental): Botulinum toxin Type A 100U injected into the detrusor, after protocol specified criteria are met, and no more frequently than every 12 weeks.
  Interventions: Biological: botulinum toxin Type A
- botulinum toxin Type A 150U (Experimental): Botulinum toxin Type A 150U injected into the detrusor, after protocol specified criteria are met, and no more frequently than every 12 weeks.
  Interventions: Biological: botulinum toxin Type A

INTERVENTIONS:
Biological: botulinum toxin Type A — Botulinum toxin Type A 100U or 150U injected into the detrusor, after protocol specified criteria are met, and no more frequently than every 12 weeks.
  Other Names: BOTOX®

SUMMARY:
The purpose of this study is to assess the long term safety and effectiveness of botulinum toxin type A in treating patients with idiopathic overactive bladder with urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Participation in preceding study 191622-095 (NCT00910845) or 191622-520 (NCT00910520)

Exclusion Criteria:

* Females who are pregnant, nursing or planning a pregnancy
* Patient has any condition or situation which, in the Investigators opinion, would put the patient at risk from continuing treatment with botulinum toxin Type A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 829 (Actual)
Dates: Start 2010-02-01 (Actual); Primary Completion 2014-08-05 (Actual); Study Completion 2014-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (8):
- Newport Beach, California, United States
- Ghent, Belgium
- Victoria, British Columbia, Canada
- Prague, Czechia
- Tübingen, Germany
- Warsaw, Poland
- Moscow, Russia
- London, United Kingdom

REFERENCES:
- [Background] Nitti VW, Ginsberg D, Sievert KD, Sussman D, Radomski S, Sand P, De Ridder D, Jenkins B, Magyar A, Chapple C; 191622-096 Investigators. Durable Efficacy and Safety of Long-Term OnabotulinumtoxinA Treatment in Patients with Overactive Bladder Syndrome: Final Results of a 3.5-Year Study. J Urol. 2016 Sep;196(3):791-800. doi: 10.1016/j.juro.2016.03.146. Epub 2016 Mar 30. PMID 27038769

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a long-term follow-up study that enrolled patients after participation in the preceding studies 191622-095 (NCT00910845) and 191622-520 (NCT00910520). A total of 829 patients received at least 1 BOTOX treatment in Study 191622-096 or in the preceding studies.
Pre-assignment Details: Following a planned interim analysis, the protocol was amended to remove the option to escalate to the 150U dose. The dose groups reflect the highest dose received (i.e. 100U BOTOX includes patients who only received 100U throughout the study and 150U BOTOX includes patients who received at least 1 dose of 150U at any time during the study).
Period: Overall Study
Arm/Group | Botulinum Toxin Type A 100U | Botulinum Toxin Type A 150U
Started | 543 | 286
Completed | 278 | 151
Not Completed | 265 | 135
Not completed — Protocol Violation | 9 | 4
Not completed — Withdrawal by Subject | 59 | 21
Not completed — Lost to Follow-up | 27 | 16
Not completed — Pregnancy | 2 | 0
Not completed — Lack of Efficacy | 15 | 32
Not completed — Adverse Event | 29 | 13
Not completed — Missing | 12 | 1
Not completed — Other Reason | 35 | 12
Not completed — Site Closed | 27 | 9
Not completed — Retreat Request >Wk 144 (exclusionary) | 4 | 5
Not completed — Study Burden | 28 | 12
Not completed — Non-Compliance | 3 | 1
Not completed — Patient Moved | 15 | 9

BASELINE CHARACTERISTICS:
Population: BOTOX-Treated population includes all patients enrolled in 191622-096 who received at least 1 BOTOX treatment in study 191622-096, 191622-095 or 191622-520. Treatment groups reflect highest dose received (100U BOTOX includes patients who received 100U throughout the study and 150U BOTOX includes patients who received at least 1 dose of 150U).
Groups:
- Total: Total of all reporting groups
Arm/Group | Botulinum Toxin Type A 100U | Botulinum Toxin Type A 150U | Total
Number analyzed (Participants) | 543 | 286 | 829
Age, Customized [Count of Participants; unit: Participants]
  <40 years | 39 | 23 | 62
  40 to 64 years | 276 | 147 | 423
  65 to 74 years | 156 | 74 | 230
  ≥75 years | 72 | 42 | 114
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 493 | 256 | 749
  Male | 50 | 30 | 80

OUTCOME MEASURES:

1. Primary Outcome: Change From Study Baseline in the Daily Average Number of Urinary Incontinence Episodes
Description: Urinary incontinence is defined as involuntary loss of urine as recorded in a patient bladder diary in the 3 consecutive days prior to each study visit for study 191622-096 (or 3 days prior to each visit in study 191622-095 or 191622-520). The number of incontinence episodes are averaged daily during this period. The initial study baseline is obtained from the patient bladder diary in the 3 consecutive days prior to the first treatment in either study 191622-095 or 191622-520. A negative number change from baseline indicates a reduction in incontinence episodes (improvement) and a positive number change from baseline indicates an increase in the number of incontinence episodes (worsening).
Time Frame: Study Baseline, Week 12 Treatment Cycle 1
Population: BOTOX-Treated Population: all patients with data at the time point who received at least 1 BOTOX treatment since the start of their clinical study participation (in study 191622-096, 191622-095 or 191622-520); analyses are based on actual treatment received
Measure: Mean (Standard Deviation); unit: Incontinence Episodes
Arm/Group | Botulinum Toxin Type A 100U
Number analyzed (Participants) | 829
Incontinence Episodes
  Study Baseline (BL) | 5.55 (3.617)
  Chg from Study BL at Wk 12 Tmt Cycle1 (N=812) | -3.26 (3.439)

2. Primary Outcome: Change From Study Baseline in the Daily Average Number of Urinary Incontinence Episodes
Description: as for outcome 1
Time Frame: Study Baseline, Week 12 Treatment Cycle 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Incontinence Episodes
Arm/Group | Botulinum Toxin Type A 100U | Botulinum Toxin Type A 150U
Number analyzed (Participants) | 608 | 116
Incontinence Episodes
  Study Baseline (BL) | 5.70 (3.685) | 5.66 (3.798)
  Chg from Study BL at Wk 12 Tmt Cycle2 (N=597, 108) | -3.64 (3.402) | -3.05 (3.690)

3. Primary Outcome: Change From Study Baseline in the Daily Average Number of Urinary Incontinence Episodes
Description: as for outcome 1
Time Frame: Study Baseline, Week 12 Treatment Cycle 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Incontinence Episodes
Arm/Group | Botulinum Toxin Type A 100U | Botulinum Toxin Type A 150U
Number analyzed (Participants) | 388 | 179
Incontinence Episodes
  Study Baseline (BL) | 5.65 (3.380) | 6.30 (4.280)
  Chg from Study BL at Wk 12 Tmt Cycle3 (N=372, 170) | -3.82 (3.341) | -3.46 (3.771)

4. Primary Outcome: Change From Study Baseline in the Daily Average Number of Urinary Incontinence Episodes
Description: as for outcome 1
Time Frame: Study Baseline, Week 12 Treatment Cycle 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Incontinence Episodes
Arm/Group | Botulinum Toxin Type A 100U | Botulinum Toxin Type A 150U
Number analyzed (Participants) | 273 | 131
Incontinence Episodes
  Study Baseline (BL) | 5.78 (3.463) | 6.19 (4.140)
  Chg from Study BL at Wk 12 Tmt Cycle4 (N=264, 122) | -3.48 (3.733) | -3.32 (3.972)

5. Primary Outcome: Change From Study Baseline in the Daily Average Number of Urinary Incontinence Episodes
Description: as for outcome 1
Time Frame: Study Baseline, Week 12 Treatment Cycle 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Incontinence Episodes
Arm/Group | Botulinum Toxin Type A 100U | Botulinum Toxin Type A 150U
Number analyzed (Participants) | 185 | 88
Incontinence Episodes
  Study Baseline (BL) | 5.47 (3.283) | 6.43 (3.622)
  Chg from Study BL at Wk 12 Tmt Cycle5 (N=181, 85) | -3.34 (3.791) | -3.58 (3.266)

6. Primary Outcome: Change From Study Baseline in the Daily Average Number of Urinary Incontinence Episodes
Description: as for outcome 1
Time Frame: Study Baseline, Week 12 Treatment Cycle 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Incontinence Episodes
Arm/Group | Botulinum Toxin Type A 100U | Botulinum Toxin Type A 150U
Number analyzed (Participants) | 139 | 50
Incontinence Episodes
  Study Baseline (BL) | 5.65 (3.238) | 7.17 (4.223)
  Chg from Study BL at Wk 12 Tmt Cycle6 (N=136, 48) | -3.05 (3.493) | -3.12 (3.753)

7. Primary Outcome: Percentage of Patients With a Positive Response on the 4-Point Treatment Benefit Scale (TBS)
Description: The TBS is a single-item scale in which the patient considers his/her current condition (urinary problems, urinary incontinence) compared with his/her condition before receiving any study treatment in study 191622-095 or 191622-520. Response options are: 1 = greatly improved; 2 = improved; 3 = not changed; and 4 = worsened. Patients scoring either "greatly improved" or "improved" are considered to have a positive response.
Time Frame: Week 12 Treatment Cycle 1
Population: as for outcome 1
Measure: Number; unit: Percentage of Patients
Arm/Group | Botulinum Toxin Type A 100U
Number analyzed (Participants) | 812
Percentage of Patients | 74.0

8. Primary Outcome: Percentage of Patients With a Positive Response on the 4-Point TBS
Description: as for outcome 7
Time Frame: Week 12 Treatment Cycle 2
Population: as for outcome 1
Measure: Number; unit: Percentage of Patients
Arm/Group | Botulinum Toxin Type A 100U | Botulinum Toxin Type A 150U
Number analyzed (Participants) | 594 | 110
Percentage of Patients | 81.3 | 71.8

9. Primary Outcome: Percentage of Patients With a Positive Response on the 4-Point TBS
Description: as for outcome 7
Time Frame: Week 12 Treatment Cycle 3
Population: as for outcome 1
Measure: Number; unit: Percentage of Patients
Arm/Group | Botulinum Toxin Type A 100U | Botulinum Toxin Type A 150U
Number analyzed (Participants) | 374 | 173
Percentage of Patients | 82.1 | 71.1

10. Primary Outcome: Percentage of Patients With a Positive Response on the 4-Point TBS
Description: as for outcome 7
Time Frame: Week 12 Treatment Cycle 4
Population: as for outcome 1
Measure: Number; unit: Percentage of Patients
Arm/Group | Botulinum Toxin Type A 100U | Botulinum Toxin Type A 150U
Number analyzed (Participants) | 263 | 123
Percentage of Patients | 78.3 | 81.3

11. Primary Outcome: Percentage of Patients With a Positive Response on the 4-Point TBS
Description: as for outcome 7
Time Frame: Week 12 Treatment Cycle 5
Population: as for outcome 1
Measure: Number; unit: Percentage of Patients
Arm/Group | Botulinum Toxin Type A 100U | Botulinum Toxin Type A 150U
Number analyzed (Participants) | 179 | 86
Percentage of Patients | 83.2 | 81.4

12. Primary Outcome: Percentage of Patients With a Positive Response on the 4-Point TBS
Description: as for outcome 7
Time Frame: Week 12 Treatment Cycle 6
Population: as for outcome 1
Measure: Number; unit: Percentage of Patients
Arm/Group | Botulinum Toxin Type A 100U | Botulinum Toxin Type A 150U
Number analyzed (Participants) | 136 | 48
Percentage of Patients | 80.9 | 81.3

13. Secondary Outcome: Change From Study Baseline in the Daily Average Number of Micturition Episodes
Description: The number of micturition (urination) episodes are recorded in a patient bladder diary in the 3 consecutive days prior to each study visit for study 191622-096 (or 3 days prior to each visit in study 191622-095 or 191622-520). The number of micturition episodes are averaged daily during this period. The initial study baseline is obtained from the patient bladder diary in the 3 consecutive days prior to the first treatment in either study 191622-095 or 191622-520. A negative number change from baseline indicates a reduction in micturition episodes (improvement) and a positive number change from baseline indicates an increase in the number of micturition episodes (worsening).
Time Frame: Study Baseline, Week 12 Treatment Cycle 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of Episodes
Arm/Group | Botulinum Toxin Type A 100U
Number analyzed (Participants) | 829
Number of Episodes
  Study Baseline (BL) | 11.70 (3.584)
  Chg from Study BL at Wk 12 Tmt Cycle1 (N=812) | -2.56 (2.887)

14. Secondary Outcome: Change From Study Baseline in the Daily Average Number of Micturition Episodes
Description: as for outcome 13
Time Frame: Study Baseline, Week 12 Treatment Cycle 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of Episodes
Arm/Group | Botulinum Toxin Type A 100U | Botulinum Toxin Type A 150U
Number analyzed (Participants) | 608 | 116
Number of Episodes
  Study Baseline (BL) | 11.83 (3.634) | 11.48 (3.912)
  Chg from Study BL at Wk 12 Tmt Cycle2 (N=597, 108) | -2.89 (3.037) | -2.31 (3.293)

15. Secondary Outcome: Change From Study Baseline in the Daily Average Number of Micturition Episodes
Description: as for outcome 13
Time Frame: Study Baseline, Week 12 Treatment Cycle 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of Episodes
Arm/Group | Botulinum Toxin Type A 100U | Botulinum Toxin Type A 150U
Number analyzed (Participants) | 388 | 179
Number of Episodes
  Study Baseline (BL) | 11.65 (3.553) | 12.22 (3.760)
  Chg from Study BL at Wk 12 Tmt Cycle3 (N=372, 170) | -2.86 (3.058) | -3.01 (3.217)

16. Secondary Outcome: Change From Study Baseline in the Daily Average Number of Micturition Episodes
Description: as for outcome 13
Time Frame: Study Baseline, Week 12 Treatment Cycle 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of Episodes
Arm/Group | Botulinum Toxin Type A 100U | Botulinum Toxin Type A 150U
Number analyzed (Participants) | 273 | 131
Number of Episodes
  Study Baseline (BL) | 11.68 (3.456) | 11.82 (3.442)
  Chg from Study BL at Wk 12 Tmt Cycle4 (N=264, 122) | -2.69 (3.485) | -2.78 (2.882)

17. Secondary Outcome: Change From Study Baseline in the Daily Average Number of Micturition Episodes
Description: as for outcome 13
Time Frame: Study Baseline, Week 12 Treatment Cycle 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of Episodes
Arm/Group | Botulinum Toxin Type A 100U | Botulinum Toxin Type A 150U
Number analyzed (Participants) | 185 | 88
Number of Episodes
  Study Baseline (BL) | 11.55 (3.261) | 11.79 (2.770)
  Chg from Study BL at Wk 12 Tmt Cycle5 (N=181, 85) | -2.85 (3.181) | -3.19 (2.772)

18. Secondary Outcome: Change From Study Baseline in the Daily Average Number of Micturition Episodes
Description: as for outcome 13
Time Frame: Study Baseline, Week 12 Treatment Cycle 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of Episodes
Arm/Group | Botulinum Toxin Type A 100U | Botulinum Toxin Type A 150U
Number analyzed (Participants) | 139 | 50
Number of Episodes
  Study Baseline (BL) | 11.85 (3.377) | 11.81 (2.990)
  Chg from Study BL at Wk 12 Tmt Cycle6 (N=136, 48) | -2.76 (3.153) | -2.66 (3.351)

19. Secondary Outcome: Change From Study Baseline in the Urinary Incontinence-Specific Quality of Life (I-QOL) Questionnaire Total Summary Score
Description: The I-QOL questionnaire is a validated, disease-specific quality of life (QOL) questionnaire containing 22 questions designed to measure the impact of urinary incontinence on patients' lives. Each question is answered on a 5-point scale (1 = worst QOL and 5 = best QOL). The scores are totaled over the 22 questions and normalized to a score of 0-100 (0 = worst QOL and 100= best QOL). The I-QOL total score is calculated by combining the 22-item subscores from the 3 I-QOL domains: Avoidance Limiting Behavior, Psychological Impact, and Social Embarrassment. The initial study baseline is obtained from data collected prior to the first treatment in Study 191622-095 or 191622-520. Positive number changes from baseline indicate improved QOL and negative changes from baseline indicate worsened QOL.
Time Frame: Study Baseline, Week 12 Treatment Cycle 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Botulinum Toxin Type A 100U
Number analyzed (Participants) | 827
Scores on a Scale
  Study Baseline (BL) | 34.3 (18.58)
  Chg from Study BL at Wk 12 Tmt Cycle1 (N=810) | 26.0 (24.84)

20. Secondary Outcome: Change From Study Baseline in the I-QOL Questionnaire Total Summary Score
Description: as for outcome 19
Time Frame: Study Baseline, Week 12 Treatment Cycle 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Botulinum Toxin Type A 100U | Botulinum Toxin Type A 150U
Number analyzed (Participants) | 606 | 116
Scores on a Scale
  Study Baseline (BL) | 33.8 (18.72) | 32.8 (17.91)
  Chg from Study BL at Wk 12 Tmt Cycle2 (N=586, 109) | 28.6 (24.38) | 21.6 (23.71)

21. Secondary Outcome: Change From Study Baseline in the I-QOL Questionnaire Total Summary Score
Description: as for outcome 19
Time Frame: Study Baseline, Week 12 Treatment Cycle 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Botulinum Toxin Type A 100U | Botulinum Toxin Type A 150U
Number analyzed (Participants) | 386 | 179
Scores on a Scale
  Study Baseline (BL) | 33.8 (18.21) | 31.9 (18.17)
  Chg from Study BL at Wk 12 Tmt Cycle3 (N=371, 173) | 27.6 (22.39) | 23.7 (25.68)

22. Secondary Outcome: Change From Study Baseline in the I-QOL Questionnaire Total Summary Score
Description: as for outcome 19
Time Frame: Study Baseline, Week 12 Treatment Cycle 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Botulinum Toxin Type A 100U | Botulinum Toxin Type A 150U
Number analyzed (Participants) | 271 | 131
Scores on a Scale
  Study Baseline (BL) | 31.4 (17.32) | 32.5 (19.36)
  Chg from Study BL at Wk 12 Tmt Cycle4 (N=261, 124) | 27.3 (24.90) | 20.3 (22.63)

23. Secondary Outcome: Change From Study Baseline in the I-QOL Questionnaire Total Summary Score
Description: as for outcome 19
Time Frame: Study Baseline, Week 12 Treatment Cycle 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Botulinum Toxin Type A 100U | Botulinum Toxin Type A 150U
Number analyzed (Participants) | 184 | 88
Scores on a Scale
  Study Baseline (BL) | 31.2 (17.49) | 31.9 (20.30)
  Chg from Study BL at Wk 12 Tmt Cycle5 (N=178, 86) | 28.1 (23.75) | 19.5 (21.43)

24. Secondary Outcome: Change From Study Baseline in the I-QOL Questionnaire Total Summary Score
Description: as for outcome 19
Time Frame: Study Baseline, Week 12 Treatment Cycle 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Botulinum Toxin Type A 100U | Botulinum Toxin Type A 150U
Number analyzed (Participants) | 138 | 50
Scores on a Scale
  Study Baseline (BL) | 30.3 (17.87) | 30.2 (20.28)
  Chg from Study BL at Wk 12 Tmt Cycle5 (N=178, 86) | 22.6 (24.99) | 18.3 (14.91)

25. Secondary Outcome: Change From Study Baseline in the King's Health Questionnaire (KHQ) Role Limitations Domain
Description: The KHQ is a disease-specific health-related QOL questionnaire that measures urinary incontinence. The role limitations domain consists of 2 questions answered on a 4-point scale (not at all, slightly, moderate, a lot). The initial study baseline is obtained from data collected prior to the first treatment in Study 191622-095 or 191622-520. Positive number changes from baseline indicate a worsening in role limitations and negative number changes from baseline indicate an improvement in role limitations.
Time Frame: Study Baseline, Week 12 Treatment Cycle 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Botulinum Toxin Type A 100U
Number analyzed (Participants) | 824
Scores on a Scale
  Study Baseline (BL) | 64.3 (28.77)
  Chg from Study BL at Wk 12 Tmt Cycle1 (N=813) | -28.5 (34.32)

26. Secondary Outcome: Change From Study Baseline in the KHQ Role Limitations Domain
Description: as for outcome 25
Time Frame: Study Baseline, Week 12 Treatment Cycle 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Botulinum Toxin Type A 100U | Botulinum Toxin Type A 150U
Number analyzed (Participants) | 605 | 115
Scores on a Scale
  Study Baseline (BL) | 64.5 (28.51) | 66.2 (30.15)
  Chg from Study BL at Wk 12 Tmt Cycle2 (N=585, 109) | -32.1 (34.29) | -29.2 (35.94)

27. Secondary Outcome: Change From Study Baseline in the KHQ Role Limitations Domain
Description: as for outcome 25
Time Frame: Study Baseline, Week 12 Treatment Cycle 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Botulinum Toxin Type A 100U | Botulinum Toxin Type A 150U
Number analyzed (Participants) | 387 | 177
Scores on a Scale
  Study Baseline (BL) | 64.7 (28.36) | 63.4 (30.41)
  Chg from Study BL at Wk 12 Tmt Cycle3 (N=373, 171) | -29.7 (33.47) | -27.9 (34.57)

28. Secondary Outcome: Change From Study Baseline in the KHQ Role Limitations Domain
Description: as for outcome 25
Time Frame: Study Baseline, Week 12 Treatment Cycle 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Botulinum Toxin Type A 100U | Botulinum Toxin Type A 150U
Number analyzed (Participants) | 272 | 130
Scores on a Scale
  Study Baseline (BL) | 66.3 (27.65) | 62.3 (31.17)
  Chg from Study BL at Wk 12 Tmt Cycle4 (N=261, 123) | -30.9 (33.82) | -23.4 (33.05)

29. Secondary Outcome: Change From Study Baseline in the KHQ Role Limitations Domain
Description: as for outcome 25
Time Frame: Study Baseline, Week 12 Treatment Cycle 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Botulinum Toxin Type A 100U | Botulinum Toxin Type A 150U
Number analyzed (Participants) | 185 | 87
Scores on a Scale
  Study Baseline (BL) | 65.4 (29.15) | 62.6 (31.84)
  Chg from Study BL at Wk 12 Tmt Cycle5 (N=179, 85) | -30.8 (35.13) | -26.3 (28.45)

30. Secondary Outcome: Change From Study Baseline in the KHQ Role Limitations Domain
Description: as for outcome 25
Time Frame: Study Baseline, Week 12 Treatment Cycle 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Botulinum Toxin Type A 100U | Botulinum Toxin Type A 150U
Number analyzed (Participants) | 138 | 50
Scores on a Scale
  Study Baseline (BL) | 66.4 (30.00) | 60.3 (33.15)
  Chg from Study BL at Wk 12 Tmt Cycle6 (N=134, 48) | -24.8 (38.93) | -22.9 (25.64)

31. Secondary Outcome: Change From Study Baseline in the KHQ Social Limitations Domain
Description: The KHQ is a disease-specific health-related QOL questionnaire that measures urinary incontinence. The social limitations domain consists of 4 questions answered on a 4-point scale (not at all, slightly, moderate, a lot). The initial study baseline is obtained from data collected prior to the first treatment in Study 191622-095 or 191622-520. Positive number changes from baseline indicate a worsening in role limitations and negative number changes from baseline indicate an improvement in role limitations.
Time Frame: Study Baseline, Week 12 Treatment Cycle 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Botulinum Toxin Type A 100U
Number analyzed (Participants) | 824
Scores on a Scale
  Study Baseline (BL) | 43.1 (30.79)
  Chg from Study BL at Wk 12 Tmt Cycle1 (N=813) | -18.4 (29.46)

32. Secondary Outcome: Change From Study Baseline in the KHQ Social Limitations Domain
Description: as for outcome 31
Time Frame: Study Baseline, Week 12 Treatment Cycle 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Botulinum Toxin Type A 100U | Botulinum Toxin Type A 150U
Number analyzed (Participants) | 605 | 115
Scores on a Scale
  Study Baseline (BL) | 43.0 (30.96) | 48.4 (30.12)
  Chg from Study BL at Wk 12 Tmt Cycle2 (N=585, 109) | -20.0 (29.12) | -19.0 (28.55)

33. Secondary Outcome: Change From Study Baseline in the KHQ Social Limitations Domain
Description: as for outcome 31
Time Frame: Study Baseline, Week 12 Treatment Cycle 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Botulinum Toxin Type A 100U | Botulinum Toxin Type A 150U
Number analyzed (Participants) | 387 | 177
Scores on a Scale
  Study Baseline (BL) | 42.8 (31.02) | 45.4 (31.38)
  Chg from Study BL at Wk 12 Tmt Cycle3 (N=373, 171) | -17.9 (29.26) | -19.2 (28.31)

34. Secondary Outcome: Change From Study Baseline in the KHQ Social Limitations Domain
Description: as for outcome 31
Time Frame: Study Baseline, Week 12 Treatment Cycle 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Botulinum Toxin Type A 100U | Botulinum Toxin Type A 150U
Number analyzed (Participants) | 272 | 130
Scores on a Scale
  Study Baseline (BL) | 44.7 (31.86) | 43.2 (30.46)
  Chg from Study BL at Wk 12 Tmt Cycle4 (N=261, 123) | -19.8 (31.26) | -16.1 (23.17)

35. Secondary Outcome: Change From Study Baseline in the KHQ Social Limitations Domain
Description: as for outcome 31
Time Frame: Study Baseline, Week 12 Treatment Cycle 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Botulinum Toxin Type A 100U | Botulinum Toxin Type A 150U
Number analyzed (Participants) | 185 | 87
Scores on a Scale
  Study Baseline (BL) | 44.4 (31.39) | 43.4 (32.89)
  Chg from Study BL at Wk 12 Tmt Cycle5 (N=179, 85) | -21.7 (28.47) | -15.7 (24.52)

36. Secondary Outcome: Change From Study Baseline in the KHQ Social Limitations Domain
Description: as for outcome 31
Time Frame: Study Baseline, Week 12 Treatment Cycle 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Botulinum Toxin Type A 100U | Botulinum Toxin Type A 150U
Number analyzed (Participants) | 138 | 50
Scores on a Scale
  Study Baseline (BL) | 46.7 (32.72) | 43.3 (32.56)
  Chg from Study BL at Wk 12 Tmt Cycle6 (N=134, 48) | -17.0 (33.59) | -17.6 (24.43)

37. Secondary Outcome: Change From Study Baseline in Daily Frequency of Urgency Episodes
Description: The number of urgency episodes are recorded in a patient bladder diary in the 3 consecutive days prior to each study visit for study 191622-096 (or 3 days prior to each visit in study 191622-095 or 191622-520). The number of urgency episodes are averaged daily during this period. The initial study baseline is obtained from the patient bladder diary in the 3 consecutive days prior to the first treatment in either study 191622-095 or 191622-520. A negative number change from baseline indicates a reduction in urgency episodes (improvement) and a positive number change from baseline indicates an increase in the number of urgency episodes (worsening).
Time Frame: Study Baseline, Week 12 Treatment Cycle 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of Episodes
Arm/Group | Botulinum Toxin Type A 100U
Number analyzed (Participants) | 829
Number of Episodes
  Study Baseline (BL) | 8.55 (4.206)
  Chg from Study BL at Wk 12 Tmt Cycle1 (N=812) | -3.81 (4.031)

38. Secondary Outcome: Change From Study Baseline in Daily Frequency of Urgency Episodes
Description: as for outcome 37
Time Frame: Study Baseline, Week 12 Treatment Cycle 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of Episodes
Arm/Group | Botulinum Toxin Type A 100U | Botulinum Toxin Type A 150U
Number analyzed (Participants) | 608 | 116
Number of Episodes
  Study Baseline (BL) | 8.63 (4.188) | 9.09 (4.764)
  Chg from Study BL at Wk 12 Tmt Cycle2 (N=597, 108) | -4.07 (4.046) | -3.96 (4.519)

39. Secondary Outcome: Change From Study Baseline in Daily Frequency of Urgency Episodes
Description: as for outcome 37
Time Frame: Study Baseline, Week 12 Treatment Cycle 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of Episodes
Arm/Group | Botulinum Toxin Type A 100U | Botulinum Toxin Type A 150U
Number analyzed (Participants) | 388 | 179
Number of Episodes
  Study Baseline (BL) | 8.62 (4.055) | 9.28 (4.552)
  Chg from Study BL at Wk 12 Tmt Cycle3 (N=372, 170) | -4.22 (4.120) | -3.86 (4.332)

40. Secondary Outcome: Change From Study Baseline in Daily Frequency of Urgency Episodes
Description: as for outcome 37
Time Frame: Study Baseline, Week 12 Treatment Cycle 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of Episodes
Arm/Group | Botulinum Toxin Type A 100U | Botulinum Toxin Type A 150U
Number analyzed (Participants) | 273 | 131
Number of Episodes
  Study Baseline (BL) | 8.65 (3.951) | 8.98 (4.241)
  Chg from Study BL at Wk 12 Tmt Cycle4 (N=264, 122) | -3.92 (4.341) | -3.50 (3.916)

41. Secondary Outcome: Change From Study Baseline in Daily Frequency of Urgency Episodes
Description: as for outcome 37
Time Frame: Study Baseline, Week 12 Treatment Cycle 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of Episodes
Arm/Group | Botulinum Toxin Type A 100U | Botulinum Toxin Type A 150U
Number analyzed (Participants) | 185 | 88
Number of Episodes
  Study Baseline (BL) | 8.67 (3.961) | 8.89 (3.341)
  Chg from Study BL at Wk 12 Tmt Cycle5 (N=181, 85) | -4.11 (4.549) | -3.56 (3.576)

42. Secondary Outcome: Change From Study Baseline in Daily Frequency of Urgency Episodes
Description: as for outcome 37
Time Frame: Study Baseline, Week 12 Treatment Cycle 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of Episodes
Arm/Group | Botulinum Toxin Type A 100U | Botulinum Toxin Type A 150U
Number analyzed (Participants) | 139 | 50
Number of Episodes
  Study Baseline (BL) | 8.98 (4.059) | 8.84 (3.629)
  Chg from Study BL at Wk 12 Tmt Cycle6 (N=136, 48) | -3.95 (4.662) | -2.64 (4.112)

ADVERSE EVENTS:
Description: BOTOX-Treated Population includes all patients who received at least 1 BOTOX treatment since the start of their clinical study participation (in study 191622-096, 191622-095 or 191622-520), and is used to assess adverse events (AEs) and serious adverse events (SAEs). AEs and SAEs are reported by treatment cycle.
Groups:
- Botulinum Toxin Type A 100U Treatment Cycle 1; Botulinum Toxin Type A 100U Treatment Cycle 2; Botulinum Toxin Type A 100U Treatment Cycle 3; Botulinum Toxin Type A 100U Treatment Cycle 4; Botulinum Toxin Type A 100U Treatment Cycle 5; Botulinum Toxin Type A 100U Treatment Cycle 6; Botulinum Toxin Type A 100U Treatment Cycle 7; Botulinum Toxin Type A 100U Treatment Cycle 8; Botulinum Toxin Type A 100U Treatment Cycle 9; Botulinum Toxin Type A 100U Treatment Cycle 10; Botulinum Toxin Type A 100U Treatment Cycle 11; Botulinum Toxin Type A 100U Treatment Cycle 12; Botulinum Toxin Type A 100U Treatment Cycle 13: Botulinum toxin Type A 100U injected into the detrusor, after protocol specified criteria are met, and no more frequently than every 12 weeks.
- Botulinum Toxin Type A 150U Treatment Cycle 2; Botulinum Toxin Type A 150U Treatment Cycle 3; Botulinum Toxin Type A 150U Treatment Cycle 4; Botulinum Toxin Type A 150U Treatment Cycle 5; Botulinum Toxin Type A 150U Treatment Cycle 6; Botulinum Toxin Type A 150U Treatment Cycle 7; Botulinum Toxin Type A 150U Treatment Cycle 8; Botulinum Toxin Type A 150U Treatment Cycle 9; Botulinum Toxin Type A 150U Treatment Cycle 10: Botulinum toxin Type A 150U injected into the detrusor, after protocol specified criteria are met, and no more frequently than every 12 weeks.
Arm/Group | Botulinum Toxin Type A 100U Treatment Cycle 1 | Botulinum Toxin Type A 100U Treatment Cycle 2 | Botulinum Toxin Type A 150U Treatment Cycle 2 | Botulinum Toxin Type A 100U Treatment Cycle 3 | Botulinum Toxin Type A 150U Treatment Cycle 3 | Botulinum Toxin Type A 100U Treatment Cycle 4 | Botulinum Toxin Type A 150U Treatment Cycle 4 | Botulinum Toxin Type A 100U Treatment Cycle 5 | Botulinum Toxin Type A 150U Treatment Cycle 5 | Botulinum Toxin Type A 100U Treatment Cycle 6 | Botulinum Toxin Type A 150U Treatment Cycle 6 | Botulinum Toxin Type A 100U Treatment Cycle 7 | Botulinum Toxin Type A 150U Treatment Cycle 7 | Botulinum Toxin Type A 100U Treatment Cycle 8 | Botulinum Toxin Type A 150U Treatment Cycle 8 | Botulinum Toxin Type A 100U Treatment Cycle 9 | Botulinum Toxin Type A 150U Treatment Cycle 9 | Botulinum Toxin Type A 100U Treatment Cycle 10 | Botulinum Toxin Type A 150U Treatment Cycle 10 | Botulinum Toxin Type A 100U Treatment Cycle 11 | Botulinum Toxin Type A 100U Treatment Cycle 12 | Botulinum Toxin Type A 100U Treatment Cycle 13
Serious Adverse Events (participants affected / at risk) | 71/829 | 62/608 | 7/116 | 32/388 | 13/179 | 18/273 | 8/131 | 15/185 | 4/88 | 8/139 | 3/50 | 3/93 | 0/27 | 4/69 | 0/11 | 0/48 | 0/7 | 1/37 | 1/2 | 2/20 | 1/5 | 0/2
Other Adverse Events (participants affected / at risk) | 297/829 | 204/608 | 28/116 | 135/388 | 50/179 | 86/273 | 34/131 | 53/185 | 35/88 | 43/139 | 10/50 | 37/93 | 16/27 | 21/69 | 9/11 | 18/48 | 6/7 | 14/37 | 1/2 | 12/20 | 1/5 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Botulinum Toxin Type A 100U Treatment Cycle 1 (N=829) | Botulinum Toxin Type A 100U Treatment Cycle 2 (N=608) | Botulinum Toxin Type A 150U Treatment Cycle 2 (N=116) | Botulinum Toxin Type A 100U Treatment Cycle 3 (N=388) | Botulinum Toxin Type A 150U Treatment Cycle 3 (N=179) | Botulinum Toxin Type A 100U Treatment Cycle 4 (N=273) | Botulinum Toxin Type A 150U Treatment Cycle 4 (N=131) | Botulinum Toxin Type A 100U Treatment Cycle 5 (N=185) | Botulinum Toxin Type A 150U Treatment Cycle 5 (N=88) | Botulinum Toxin Type A 100U Treatment Cycle 6 (N=139) | Botulinum Toxin Type A 150U Treatment Cycle 6 (N=50) | Botulinum Toxin Type A 100U Treatment Cycle 7 (N=93) | Botulinum Toxin Type A 150U Treatment Cycle 7 (N=27) | Botulinum Toxin Type A 100U Treatment Cycle 8 (N=69) | Botulinum Toxin Type A 150U Treatment Cycle 8 (N=11) | Botulinum Toxin Type A 100U Treatment Cycle 9 (N=48) | Botulinum Toxin Type A 150U Treatment Cycle 9 (N=7) | Botulinum Toxin Type A 100U Treatment Cycle 10 (N=37) | Botulinum Toxin Type A 150U Treatment Cycle 10 (N=2) | Botulinum Toxin Type A 100U Treatment Cycle 11 (N=20) | Botulinum Toxin Type A 100U Treatment Cycle 12 (N=5) | Botulinum Toxin Type A 100U Treatment Cycle 13 (N=2)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Supraventricular Tachycardia (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angina Pectoris (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 2 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac Failure Congestive (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coronary Artery Disease (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Crohn's Disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inguinal Hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Volvulus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foramen Magnum Stenosis (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 2 | 0 | 3 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Appendiceal Abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis Viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Comminuted Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metabolic Acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 | 8 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Foot Deformity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 5 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast Cancer Stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung Carcinoma Cell Type Unspecified Stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/80 | 0/55 | 0/15 | 0/26 | 0/15 | 0/16 | 0/8 | 0/13 | 0/5 | 0/7 | 0/1 | 0/5 | 0/1 | 0/3 | 0/1 | 0/2 | 0/1 | 0/3 | 0/0 | 0/2 | 0/1 | 0/0 — MALE ONLY
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/749 | 0/553 | 0/101 | 0/362 | 0/164 | 0/257 | 0/123 | 0/172 | 0/83 | 0/132 | 0/49 | 0/88 | 0/26 | 0/66 | 0/10 | 0/46 | 0/6 | 0/34 | 0 | 0/18 | 0/4 | 0 — FEMALE ONLY
Bulbar Palsy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Carpal Tunnel Syndrome (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Major Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal Failure Acute (Renal and urinary disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary Retention (Renal and urinary disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Calculus Ureteric (Renal and urinary disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urge Incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1/80 | 0/55 | 0/15 | 0/26 | 0/15 | 0/16 | 0/8 | 0/13 | 1/5 | 0/7 | 0/1 | 0/5 | 0/1 | 0/3 | 0/1 | 0/2 | 0/1 | 0/3 | 0/0 | 0/2 | 0/1 | 0/0 — MALE ONLY
Polycystic Ovaries (Reproductive system and breast disorders) | 1/749 | 0/553 | 0/101 | 0/362 | 0/164 | 0/257 | 0/123 | 0/172 | 0/83 | 0/132 | 0/49 | 0/88 | 0/26 | 0/66 | 0/10 | 0/46 | 0/6 | 0/34 | 0 | 0/18 | 0/4 | 0 — FEMALE ONLY
Uterine Haemorrhage (Reproductive system and breast disorders) | 1/749 | 1/553 | 0/101 | 0/362 | 0/164 | 0/257 | 0/123 | 0/172 | 0/83 | 0/132 | 0/49 | 0/88 | 0/26 | 0/66 | 0/10 | 0/46 | 0/6 | 0/34 | 0 | 0/18 | 0/4 | 0 — FEMALE ONLY
Vaginal Prolapse (Reproductive system and breast disorders) | 1/749 | 1/553 | 0/101 | 0/362 | 0/164 | 0/257 | 0/123 | 0/172 | 0/83 | 0/132 | 0/49 | 0/88 | 0/26 | 0/66 | 0/10 | 0/46 | 0/6 | 0/34 | 0 | 0/18 | 0/4 | 0 — FEMALE ONLY
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Preventive Surgery (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arterial Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Internal Hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large Intestine Polyp (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hernia Obstructive (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Medical Device Complication (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 3 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infected Skin Ulcer (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint Dislocation (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Patella Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stress Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tibia Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sigmoidoscopy (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Benign Neoplasm of Spinal Cord (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thyroid Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral Infarction (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular Disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Obturator Neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Restless Legs Syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage Intracranial (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression Suicidal (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Suicide Attempt (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis Interstitial (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cervical Polyp (Reproductive system and breast disorders) | 0/749 | 1/553 | 0/101 | 0/362 | 0/164 | 0/257 | 0/123 | 0/172 | 0/83 | 0/132 | 0/49 | 0/88 | 0/26 | 0/66 | 0/10 | 0/46 | 0/6 | 0/34 | 0 | 0/18 | 0/4 | 0 — FEMALE ONLY
Uterine Prolapse (Reproductive system and breast disorders) | 0/749 | 1/553 | 0/101 | 1/362 | 0/164 | 0/257 | 0/123 | 0/172 | 0/83 | 0/132 | 0/49 | 0/88 | 0/26 | 0/66 | 0/10 | 0/46 | 0/6 | 0/34 | 0 | 0/18 | 0/4 | 0 — FEMALE ONLY
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Swelling Face (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arterial Occlusive Disease (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angina Unstable (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stress Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Congenital Diaphragmatic Hernia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device Ineffective (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Allergy to Plants (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaphylactic Shock (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacterial Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Accidental Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Incisional Hernia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyogenic Granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Benign Ovarian Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/749 | 0/553 | 0/101 | 0/362 | 1/164 | 0/257 | 0/123 | 0/172 | 0/83 | 0/132 | 0/49 | 0/88 | 0/26 | 0/66 | 0/10 | 0/46 | 0/6 | 0/34 | 0 | 0/18 | 0/4 | 0 — FEMALE ONLY
Lip Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Carotid Artery Stenosis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral Artery Thrombosis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cervical Radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Parkinsonism (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peroneal Nerve Palsy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transient Ischaemic Attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mental Status Changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hydroureter (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvi-Ureteric Obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0/749 | 0/553 | 0/101 | 1/362 | 0/164 | 0/257 | 0/123 | 0/172 | 0/83 | 0/132 | 0/49 | 0/88 | 0/26 | 0/66 | 0/10 | 0/46 | 0/6 | 0/34 | 0 | 0/18 | 0/4 | 0 — FEMALE ONLY
Perineal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arterial Disorder (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Temporal Arteritis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Varicose Vein (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitreous Floaters (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound Dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendon Disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant Melanoma in Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
B-Cell Small Lymphocytic Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Excessive skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertensive Crisis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mitral Valve Prolapse (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Goitre (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterovesical Fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Forearm Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Heart Rate Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional State (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Endometrial Hypertrophy (Reproductive system and breast disorders) | 0/749 | 0/553 | 0/101 | 0/362 | 0/164 | 0/257 | 0/123 | 0/172 | 1/83 | 0/132 | 0/49 | 0/88 | 0/26 | 0/66 | 0/10 | 0/46 | 0/6 | 0/34 | 0 | 0/18 | 0/4 | 0 — FEMALE ONLY
Arthritis Bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glomerulonephritis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous Cell Carcinoma of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Radiation Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin Wrinkling (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac Arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Botulinum Toxin Type A 100U Treatment Cycle 1 (N=829) | Botulinum Toxin Type A 100U Treatment Cycle 2 (N=608) | Botulinum Toxin Type A 150U Treatment Cycle 2 (N=116) | Botulinum Toxin Type A 100U Treatment Cycle 3 (N=388) | Botulinum Toxin Type A 150U Treatment Cycle 3 (N=179) | Botulinum Toxin Type A 100U Treatment Cycle 4 (N=273) | Botulinum Toxin Type A 150U Treatment Cycle 4 (N=131) | Botulinum Toxin Type A 100U Treatment Cycle 5 (N=185) | Botulinum Toxin Type A 150U Treatment Cycle 5 (N=88) | Botulinum Toxin Type A 100U Treatment Cycle 6 (N=139) | Botulinum Toxin Type A 150U Treatment Cycle 6 (N=50) | Botulinum Toxin Type A 100U Treatment Cycle 7 (N=93) | Botulinum Toxin Type A 150U Treatment Cycle 7 (N=27) | Botulinum Toxin Type A 100U Treatment Cycle 8 (N=69) | Botulinum Toxin Type A 150U Treatment Cycle 8 (N=11) | Botulinum Toxin Type A 100U Treatment Cycle 9 (N=48) | Botulinum Toxin Type A 150U Treatment Cycle 9 (N=7) | Botulinum Toxin Type A 100U Treatment Cycle 10 (N=37) | Botulinum Toxin Type A 150U Treatment Cycle 10 (N=2) | Botulinum Toxin Type A 100U Treatment Cycle 11 (N=20) | Botulinum Toxin Type A 100U Treatment Cycle 12 (N=5) | Botulinum Toxin Type A 100U Treatment Cycle 13 (N=2)
Urinary Tract Infection (Infections and infestations) | 225 | 161 | 17 | 107 | 39 | 67 | 28 | 40 | 20 | 28 | 6 | 24 | 4 | 9 | 3 | 13 | 2 | 9 | 1 | 4 | 0 | 1
Bacteriuria (Infections and infestations) | 70 | 54 | 8 | 32 | 5 | 21 | 5 | 11 | 7 | 10 | 2 | 8 | 2 | 4 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Dysuria (Renal and urinary disorders) | 71 | 47 | 7 | 20 | 16 | 15 | 8 | 7 | 9 | 9 | 3 | 6 | 5 | 1 | 2 | 3 | 0 | 1 | 0 | 0 | 0 | 1
Erectile Dysfunction (Reproductive system and breast disorders) | 0/180 | 1/55 | 0/15 | 0/26 | 1/15 | 0/16 | 0/8 | 0/13 | 0/5 | 0/7 | 0/1 | 0/5 | 0/1 | 0/3 | 0/1 | 0/2 | 0/1 | 0/3 | 0/0 | 0/2 | 0/1 | 0/0 — MALE ONLY
Depression (Psychiatric disorders) | 14 | 9 | 1 | 7 | 4 | 3 | 2 | 2 | 5 | 2 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1/80 | 0/55 | 0/15 | 0/26 | 0/15 | 0/16 | 0/8 | 0/13 | 1/5 | 0/7 | 0/1 | 0/5 | 0/1 | 0/3 | 0/1 | 0/2 | 0/1 | 0/3 | 0/0 | 0/2 | 0/1 | 0/0 — MALE ONLY
Diarrhoea (Gastrointestinal disorders) | 23 | 20 | 2 | 5 | 4 | 6 | 4 | 4 | 2 | 2 | 2 | 1 | 3 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 8 | 8 | 2 | 1 | 1 | 2 | 2 | 1 | 2 | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 26 | 19 | 2 | 11 | 4 | 5 | 0 | 4 | 0 | 3 | 0 | 2 | 2 | 2 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 12 | 6 | 4 | 12 | 2 | 2 | 1 | 3 | 2 | 3 | 0 | 1 | 2 | 1 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 27 | 26 | 1 | 8 | 3 | 6 | 4 | 3 | 2 | 2 | 1 | 1 | 2 | 5 | 1 | 2 | 0 | 1 | 0 | 2 | 0 | 0
Cataract (Eye disorders) | 8 | 8 | 0 | 7 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 13 | 14 | 0 | 2 | 2 | 3 | 2 | 2 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 30 | 17 | 5 | 7 | 5 | 5 | 5 | 6 | 2 | 2 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 13 | 23 | 5 | 13 | 4 | 2 | 1 | 7 | 3 | 2 | 2 | 1 | 0 | 1 | 1 | 4 | 1 | 0 | 0 | 0 | 0 | 0
Acute Sinusitis (Infections and infestations) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 21 | 1 | 9 | 6 | 4 | 3 | 2 | 0 | 3 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 13 | 16 | 1 | 6 | 0 | 3 | 0 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 8 | 5 | 0 | 4 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis Glandularis (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 20 | 1 | 6 | 2 | 1 | 1 | 3 | 0 | 2 | 2 | 0 | 0 | 4 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 5 | 7 | 0 | 3 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Swelling Face (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye Inflammation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 24 | 14 | 2 | 11 | 1 | 7 | 1 | 4 | 2 | 4 | 2 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Respiratory Tract Infection (Infections and infestations) | 2 | 2 | 0 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Limb Injury (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Benign Neoplasm of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 10 | 13 | 3 | 6 | 4 | 1 | 2 | 1 | 1 | 2 | 2 | 2 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Urinary Retention (Renal and urinary disorders) | 34 | 23 | 0 | 11 | 4 | 7 | 2 | 3 | 3 | 3 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0
Skin Wrinkling (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Radiation Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 3 | 2 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 3 | 9 | 0 | 3 | 1 | 2 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 6 | 3 | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 25 | 12 | 2 | 8 | 2 | 2 | 2 | 3 | 2 | 4 | 0 | 4 | 1 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Urinary Incontinence (Renal and urinary disorders) | 4 | 4 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 3 | 4 | 0 | 2 | 0 | 2 | 2 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 3 | 3 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Capsular Contracture Associated with Breast Implant (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 8 | 7 | 0 | 3 | 3 | 1 | 2 | 1 | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 3 | 4 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 4 | 2 | 1 | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Residual Urine Volume (Investigations) | 26 | 12 | 0 | 10 | 2 | 4 | 2 | 2 | 1 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Trigeminal Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Psychotic Disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bladder Hypertrophy (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urine Abnormality (Renal and urinary disorders) | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 5 | 4 | 0 | 6 | 1 | 3 | 0 | 2 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hand Fracture (Injury, poisoning and procedural complications) | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cervical Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.